CLINICAL TRIAL: NCT04851561
Title: Risk Factors for Post-coronavirus Disease-2019 Fatigue: a Prospective Case-control Study
Brief Title: Post-coronavirus Disease-2019 Fatigue
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RMC-0834-20
Record Dates: First submitted 2021-04-11; First posted 2021-04-20 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Post-COVID / Long-COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Adults recovered from COVID-19 (diagnosed using a polymerase chain reaction test from a nasopharyngeal sample), cases will be defined as such if fulfill for the following criteria: individuals who report on lasting fatigue symptoms which appeared following COVID-19, while at least two months have elapsed since COVID-19 diagnosis and the lasting fatigue symptoms are present for at least six weeks.
  Interventions: Diagnostic Test: Cardiopulmonary stress test (CPET)
- Controls: Adults recovered from COVID-19 (diagnosed using a polymerase chain reaction test from a nasopharyngeal sample), did not report fatigue symptoms at any time point following their diagnosis with COVID-19.
  Interventions: Diagnostic Test: Cardiopulmonary stress test (CPET)

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary stress test (CPET) — Cardiopulmonary stress test will be conducted under the guidance of sports and exercise physicians and nursing staff. Electrocardiogram, spirometry, blood pressure and gas exchange measuring will be assessed at rest. The participants will then undergo CPET according to a modified Astrand treadmill test protocol. The test will be terminated at maximal exercise or upon the appearance of limiting symptoms. Continuous electrocardiogram and repeated blood pressure measuring will be conducted at the recovery phase. Post-exercise spirometry will also be assessed.
  Other Names: Blood sampling

SUMMARY:
Background: COVID-19 is consistently spreading throughout the world, and the number of recovered patients is steadily increasing. Accordingly, a significant number of individuals will develop persisting post-COVID symptoms, while many of them will report on lasting fatigue. The main objective of the current study is to assess risk factors for the development of post-COVID-19 fatigue symptoms. As a secondary aim, the current study is intended to identify pathophysiology and explanatory mechanisms for the post-COVID-19 fatigue.

Study design and population: a nested case-control study will be conducted at Rabin Medical Center (RMC), Beilinson Hospital. RMC runs a post-COVID-19 clinic for adult (age ≥18 years) recovered individuals (diagnosed using a polymerase chain reaction test from a nasopharyngeal sample), who are invited for a comprehensive medical evaluation. During a visit, all individuals undergo pulmonary function testing and an evaluation by an infectious diseases physician, a pulmonologist, and a social worker. The cohort of recovered COVID-19 individuals evaluated at RMC will serve as the population from which the current study participants will be consecutively sampled. The cases would be defined as such if report on lasting fatigue symptoms which appeared following COVID-19, while at least two months have elapsed since COVID-19 diagnosis and the lasting fatigue symptoms are present for at least six weeks. The controls would be defined as those that did not report on fatigue symptoms at any time point since one month following their diagnosis with COVID-19.

Evaluation protocol of cases and controls: All participating individuals (cases and controls) will be assessed following the study protocol. The assessment will be conducted as follows:

First assessment meeting (approximately one hour long) in which the participant will undergo physical examination and blood tests, fill the study questionnaires [demographic, clinical and post-COVID fatigue questionnaire; sleep assessment questionnaires (Epworth sleepiness score [ESS], Pittsburg sleep quality index [PSQI], Insomnia severity index (ISI)]) and depression severity questionnaire (the patient health questionnaire-9 [PHQ-9]), and conduct cognitive fatigue task.

Second assessment meeting: (approximately one hour long) in which the participants will undergo a cardiopulmonary stress test (CPET).

Data collection: The main dependent variable will be the presence of continuing fatigue symptoms. The independent variables included demographic and clinical characteristics. The demographic variables will include: age at diagnosis, sex, marital status and number of children, occupational status (employed, unemployed, or retired), education (number of years at school and higher education), and occupation. The clinical variables will include: smoking status, alcohol and cannabis consumption, basic physical function (independent, limited in certain activities, dependent in activities of daily living, or bedridden), background illnesses, and pharmacotherapy. The acute COVID-19 history will be also collected: disease severity according to the WHO criteria, symptoms (sore throat, nasal congestion, headache anosmia/disguesia, cough, shortness of breath, chest pain, gastrointestinal symptoms, and myalgia), need for hospitalization, hospital complications (veno-thromboembolism, super-imposed bacterial infections), for individuals who were not hospitalized - the site of isolation (home, hotel or another isolation facility) will be collected, time from onset to symptoms resolution, pharmacotherapy directed at COVID-19, and information of other household or family members who were also diagnosed.

Statistical methods: Demographic and clinical variables of the patients with fatigue symptoms (cases) and control group (free from fatigue symptoms) will be compared using bivariate and multivariable conditional logistic regression models. Independent variables will be selected to be included in the multivariable model based on the bivariate analysis. Odds ratios and 95% confidence intervals will be obtained from the conditional logistic regression models. P<0.05 will be considered statistically significant.

Sample size calculation: Disease severity may serve as a potential risk factor for the development of lasting fatigue symptoms. A preliminary analysis revealed that in our cohort of recovered COVID-19 patients, 20% were hospitalized due to their disease's severity. We will therefore assume that the proportions of individuals required hospitalization during the acute phase were 30% and 10% of the cases and controls, respectively. It is also likely that approximately two thirds of our sample would report on persisting fatigue. Under these assumptions, a sample size of 153 individuals (102 in the cases group and 51 in the control group) will yield a statistical power of 80% at a significance level of 5% for detecting a difference of 0.2 between two proportions.

DETAILED DESCRIPTION:
The evaluation of both cases and controls will include the following:

* Physical examination: a comprehensive physical examination, including neurological assessment of motor function.
* Blood tests: complete blood count, C-reactive protein, erythrocyte sedimentation rate, thyroid functions (TSH, fT3, fT4), kidney and liver functions, creatine phosphokinase, serum electrolytes, Epstein-Barr virus and cytomegalovirus serology testing, ferritin, and serum vitamin B12 and folate levels.
* Sleep assessment: in order to estimate the quality and characteristics of sleep, the participating individuals will independently fill the following sleep assessment questionnaires:

  * Epworth sleepiness score (ESS) - to generally evaluate subjective sleepiness (was validated in Hebrew).
  * Pittsburg sleep quality index (PSQI) - to evaluate the quality of sleep (was validated in Hebrew).
  * Insomnia severity index (ISI) - to evaluate insomnia (a Hebrew version exists, but the questionnaire is yet to be validated).
* Depression severity questionnaire: in order to screen for depression and to estimate the degree of depression severity, the participating individuals will independently fill the patient health questionnaire-9 (PHQ-9).
* Fatigue classification tool

For chronic fatigue syndrome, the Centers for Disease Control and Prevention (CDC) adopted the clinical case definition suggested by the Institute of Medicine (IOM), and consolidated criteria. We adopted the portion on fatigue from the CDC criteria for chronic fatigue syndrome, and modified it to suit for the time frame and relations with COVID-19:

Patient has a substantial reduction or impairment in the ability to engage in pre-illness levels of occupational, educational, social, or personal activities that persists for >6 weeks and is accompanied by fatigue, which is often profound, is of new onset (appeared after the diagnosis of COVID-19), is not the result of ongoing excessive exertion, and is not substantially alleviated by rest. These symptoms are present at least half of the day time, to at least a moderately severe degree.

Each participant will independently fill a designated form in which the aforementioned criteria will be mentioned, followed by to statement from which the participant will circle the one relevant for him:

* The criteria above accurately describe my current situation.
* The criteria above do not accurately reflect my current situation.

  * Assessment of exercise physiology: All participants will undergo a cardiopulmonary stress test (CPET), under the guidance of sports and exercise physicians and nursing staff. Electrocardiogram, spirometry, blood pressure and gas exchange measuring will be assessed at rest. The participants will then undergo CPET according to a modified Astrand treadmill test protocol. The test will be terminated at maximal exercise or upon the appearance of limiting symptoms . Continuous electrocardiogram and repeated blood pressure measuring will be conducted at the recovery phase. Post-exercise spirometry will also be assessed.
  * Assessment of cognitive fatigue: in order to assess cognitive fatigue, all participants will undergo the visual vigilance test. This test, that was designed to be a measure of sustained attention, was previously implemented in individuals with multiple sclerosis. This test will be conducted in a designated room in which the participants will seat in front of a computer, and will independently conduct the task after being instructed by the primary investigator or one of the sub-investigators. During the task, the different alphabetical letters will be screened at a rate of 500 milliseconds per each. The tested individual will be instructed to press the space button whenever two specific letters (i.e. the target letters) are presented. A total of 600 letters will be screened, of which 120 will be the target letters. The test is to be repeated 3 times, 5 minutes for each run. The percentage of correct presses, the number of errors and the mean reaction time will be evaluated for each time period.

ELIGIBILITY:
Inclusion Criteria:

• Adult individuals (age ≥18 years) recovered from COVID-19 (diagnosed using a polymerase chain reaction test from a nasopharyngeal sample), with or without lasting fatigue symptoms, which appeared following COVID-19, while at least two months have elapsed since COVID-19 diagnosis.

Exclusion Criteria:

* Individuals hospitalized in intensive care unit and/or required mechanical ventilation during their acute illness.
* Individuals diagnosed with pulmonary veno-thromboembolism/pulmonary infarction, on current oxygen supplementation, with sleep apnea/hypopnea syndrome or with post-COVID-19 chest imaging suggesting pulmonary fibrosis.
* Individuals with heart failure, acute coronary syndrome or percutaneous cardiac intervention during the year prior to the diagnosis.
* Individuals who underwent surgical procedure under general anesthesia during the year prior to the diagnosis.
* Individuals with cerebrovascular disease and a history of cerebrovascular accident or transient ischemic attack.
* Individuals with paralysis of the lower limbs, amputees, bedridden, those assisted with walking aids or wheelchair.
* Individuals with myopathies or myositis, degenerative neurological or muscular diseases, and myasthenia gravis.
* Individuals with pre-COVID-19 diagnosis of chronic fatigue syndrome, fibromyalgia, major depressive disorder, obstructive sleep hypopnea/apnea syndrome, or sleep disturbance necessitating pharmacotherapy.
* Individuals with chronic illnesses (autoimmune diseases and malignancies) necessitating immunosuppression (including corticosteroid therapy) or immunomodulation (including anti-cancer agents).
* Individuals with thyroid dysfunction prior to their diagnosis with COVID-19: uncontrolled hypothyroidism or hyperthyroidism and those with imbalanced thyroid stimulating hormone (TSH) level.
* Pregnant women.
* Individuals with chronic use of opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals evaluated at Rabin Medical Center's post-COVID-19 clinic for recovered adult individuals.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Pathological CPET | Up to 6 weeks from recruitment and initial testing to CPET testing
  An abnormal CPET due to either decreased respiratory capacity, muscle weakness or deconditioning

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Derived] Margalit I, Yelin D, Sagi M, Rahat MM, Sheena L, Mizrahi N, Gordin Y, Agmon H, Epstein NK, Atamna A, Tishler O, Daitch V, Babich T, Abecasis D, Yarom Y, Kazum S, Shitenberg D, Baltaxe E, Elkana O, Shapira-Lichter I, Leibovici L, Yahav D. Risk Factors and Multidimensional Assessment of Long Coronavirus Disease Fatigue: A Nested Case-Control Study. Clin Infect Dis. 2022 Nov 14;75(10):1688-1697. doi: 10.1093/cid/ciac283. PMID 35403679